CLINICAL TRIAL: NCT06533618
Title: Characterization of the "Transfusion-dependent Prediabetes" Using Continuous Glucose Monitoring: the Hemoglycare Study
Brief Title: Characterization of the "Transfusion-dependent Prediabetes" Using Continuous Glucose Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Angela Zanfardino, Medical Doctor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Hemoglycare
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Thalassemic patients (Experimental): Patient affected by TDD
  Interventions: Diagnostic Test: Continuous glucose monitoring system
- Healthy controls (Experimental): caucasian; age ≥18 years; body mass index <25.0 kg/m2; no chronic illness or medications that might affect glucose metabolism; fasting glycemia<100 mg/dl; HbA1c <5.7% (39 mmol/mol); no positive islet autoantibodies; HOMA-IR <2.5
  Interventions: Diagnostic Test: Continuous glucose monitoring system
- Euglycemic thalassemic patients (Experimental): Glucose metrics characteristic: (Time above range≥140 mg/dl: ≤ 6%)
  Interventions: Diagnostic Test: Continuous glucose monitoring system
- Hyperglicemic thalassemic patients (Experimental): Glucose metrics characteristic: (Time above range≥140 mg/dl: >6%)
  Interventions: Diagnostic Test: Continuous glucose monitoring system

INTERVENTIONS:
Diagnostic Test: Continuous glucose monitoring system — All participants (subjects and controls) applied a Medtronic Guardian4 sensor for seven days.

SUMMARY:
Dysglycemia is a frequent finding in transfusion-dependent thalassemia (TDT). The oral glucose tolerance test (OGTT) remains the only validated screening test, but the procedure is complex and time-consuming. Continuous glucose monitoring (CGM) systems are simple to use, and could have a role in the diabetes mellitus diagnosis. This study involved 39 participants (19 cases and 20 healthy controls) using CGM for the analysis of the glucose metrics. Participants resulted negative for diabetes mellitus screening tests. Patients' clinical data were compared with glucose metrics.

DETAILED DESCRIPTION:
The selection of patients took place randomly among adult patients suffering from transfusion-dependent thalassemia (TDT) belonging to the Pediatric Hematology and Oncology Unit of the AOU University of Campania "L. Vanvitelli". Patients had a history of at least 10 years of therapy with red blood cell transfusions (transfusion frequency less than one months) and iron chelation therapy. Cases tested negative for diabetes mellitus screening tests (fasting glycemia, OGTT).

Some healthy volunteers were also recruited among medical resident and doctors. Major eligibility criteria for the volunteers were: caucasian; age ≥18 years; body mass index <25.0 kg/m2; no chronic illness or medications that might affect glucose metabolism; fasting glycemia<100 mg/dl; HbA1c <5.7% (39 mmol/mol); no positive islet autoantibodies; HOMA-IR <2.5. Female participants pregnant at the time of study enrollment were not eligible.

All procedures performed in this study were approved by the Institutional Research Committee of the University of Campania "Luigi Vanvitelli". All participants have provided written consent.

Demographic and Clinical characteristics A brief schedule was specifically designed and completed by clinicians (diabetologists or hematologists) to record demographic and clinical data, including age, gender, height, weight, duration of illness, and other medical conditions (family history of diabetes, endocrine disorders, cigarette smoking habit). Finally, the HOMA-IR was calculated as a parameter for evaluating insulin resistance. Possible missing data was obtained by reviewing medical charts

Study design

All participants (subjects and controls) applied a Medtronic Guardian4 sensor for seven days. At the end of the monitoring, the glucose sensor data was analyzed using the Carelink System software.

Glucose metrics considered for the analysis were glucose management indicator (GMI), mean glucose (mg/dl), glycemic variability as standard deviation (SD) and coefficient of variation (CV), time spent with glycemia greater than or equal to 200 mg /dl (TAR200%,median), time spent with blood glucose greater than or equal to 140 mg/dl (TAR140%, median), time spent with blood glucose less than 70 mg/dl (TBR<70%, median).

As it is described in the American Diabetes Association (ADA) guidelines ,2h-glucose value ≥ 140 mg/dl (7.8 mmol/L) and <199 mg/dl (11 mmol/l) during OGTT is diagnostic for prediabetes. Moreover, 2h glucose value ≥200 mg/dl(11.1 mmol/L) during OGTT or a random glucose value (in any time of the day without regard to time since previous meal) ≥200 mg/dl(11.1 mmol/L) are both diagnostic for diabetes mellitus.

During a continuous glucose monitoring (CGM) it is not easy to understand correlation between glucose values and meals. Furthermore, in this study, the evaluation of glucose values (during CGM) two hours after a controlled meal (75-g of oral glucose in OGTT) was not performed. Instead, the participants' glucose values were observed in real life. Therefore, although the number of participants who exceeded or equaled the value 140 mg/dl or the value 200mg/dl was recorded, in addition how long these patients remained with glucose values above these cut-offs (TAR140%; TAR200%)was registered, to make the observation of abnormal glycemic profiles more precise.

Finally, the value ≤6% of TAR 140%was used as an index of normality (as indicated in other studies on healthy volunteers).

ELIGIBILITY:
Inclusion Criteria:

* They were affected by transfusion-dependent thalassemia (TDT)
* They had a history of at least 10 years of therapy with red blood cell transfusions (transfusion frequency less than one months) and iron chelation therapy
* They tested negative for diabetes mellitus screening tests (fasting glycemia, OGTT).

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with pre diabetes in Transfusion dependent patients | Seven days
  Transfusion dependent patients were studied using a continuous glucose monitoring system with the aim to show condition of dysglicemia (prediabetes)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Zanfardino, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Centro di Diabetologia Pediatrica "G.Stoppoloni", Naples, Italy

IPD SHARING:
Plan to Share IPD: No
We could share our data via a shared folder in the cloud

REFERENCES:
- [Background] Naberezhnykh GA, Khomenko VA, Krasikova IN, Kim NIu, Solov'eva TF. [Cooperative interaction between protein-porin and lipopolysaccharide]. Bioorg Khim. 1996 Sep;22(9):671-7. Russian. PMID 8999784
- [Background] De Sanctis V, Soliman A, Yassin M. Iron overload and glucose metabolism in subjects with beta-thalassaemia major: an overview. Curr Diabetes Rev. 2013 Jul;9(4):332-41. doi: 10.2174/1573399811309040005. PMID 23687960
- [Background] Karlen A, Johansson AM, Kenne L, Arvidsson LE, Hacksell U. Conformational analysis of the dopamine-receptor agonist 5-hydroxy-2-(dipropylamino)tetralin and its C(2)-methyl-substituted derivative. J Med Chem. 1986 Jun;29(6):917-24. doi: 10.1021/jm00156a008. PMID 3712382
- [Background] Miller E, Polonsky WH, Miller K. What Role Might There Be for Continuous Glucose Monitoring in the Assessment of Diabetes Risk? Diabetes Technol Ther. 2023 Jun;25(S3):S14-S20. doi: 10.1089/dia.2023.0136. PMID 37306445